CLINICAL TRIAL: NCT04255498
Title: Understanding Gulf War Illness: An Integrative Modeling Approach
Brief Title: Understanding GWI: Integrative Modeling
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Florida Veterans Affairs Foundation for Research and Education (U.S. Federal Agency)
Collaborators: Nova Southeastern University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Klimas, Director, Environmental Medicine Research and Clinical Program, South Florida Veterans Affairs Foundation for Research and Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4987.84
Record Dates: First submitted 2018-08-24; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Gulf War Illness; Persian Gulf Syndrome; Occupational Diseases
Keywords: Anti-neuroinflammatory; Homeostatic regulation; HPA axis regulator
MeSH Terms: conditions — Persian Gulf Syndrome; Occupational Diseases | interventions — Etanercept; Mifepristone

STUDY DESIGN:
Intervention Model Description: Perform Phase I study of etanercept (50 mg, once a week for 4 weeks), followed by mifepristone (300 mg, once a day for 7 days), followed by a 10 week observation period and assessment of safety, efficacy and biomarker response to therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etanercept (Experimental): 50 MG/ML Prefilled Syringe (once a week for 4 weeks)
  Interventions: Drug: Etanercept
- Mifepristone (Experimental): (300 mg once a day for 7 days) will follow the etanercept.
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Etanercept — Perform Phase I study of etanercept (50 mg, once a week for 4 weeks), followed by mifepristone (300 mg, once a day for 7 days), followed by a 10 week observation period and assessment of safety, efficacy and biomarker response to therapy.
  Perform dynamic modeling studies before and after 5 weeks of therapy, repeating the method used previously, in order to document the response to exercise and better quantify the degree of recovery in treated subjects using an exercise challenge and 9 point in time with blood and saliva collections over 24 hours with genomic, cytokine, neuropeptide and cell population studies.
  Other Names: Enbrel
  Arms: Etanercept
Drug: Mifepristone — Perform Phase I study of etanercept (50 mg, once a week for 4 weeks), followed by mifepristone (300 mg, once a day for 7 days), followed by a 10 week observation period and assessment of safety, efficacy and biomarker response to therapy.
  Perform dynamic modeling studies before and after 5 weeks of therapy, repeating the method used previously, in order to document the response to exercise and better quantify the degree of recovery in treated subjects using an exercise challenge and 9 point in time with blood and saliva collections over 24 hours with genomic, cytokine, neuropeptide and cell population studies.
  Other Names: Mifeprex
  Arms: Mifepristone

SUMMARY:
The investigator proposes to perform a Phase I study assessing safety, efficacy, and biomarker response to the therapeutic interventions of Etanercept followed by mifepristone for veterans with Gulf War Illness. The investigator will conduct and repeat the exercise challenge before treatment and on therapy to assess the impact of the interventions on homeostatic regulation and the dynamic model identified in prior studies.

DETAILED DESCRIPTION:
In the Investigator's prior work, the investigator used an exercise stress model (rest, peak oxygen consumption oxygen uptake, and 7 follow-up sampling points) to measure the mediators of relapse in the context of their interactive homeostatic networks. The investigator surveyed the response of genes and blood-borne biomarkers in order to interrogate and map the regulation of neuro-endocrine-autonomic-immune function in these subjects as compared to GW era sedentary healthy controls. This study is the first to test in the GWI human system of the impact of interventions that hope to permanently re-set the key pathway(s) involved in maintaining a "sick" homeostatic network in Gulf War Illness, discovered in our prior CDMRP and VA funded projects. An open-label Phase I study will be performed with Etanercept (once a week for 4 weeks) followed by mifepristone (once a day for 7 days), followed by a 10-week observation to assess safety, efficacy and biomarker response to maximal exercise. The impact of the interventions will be measured on current computational modeling of dynamic response GWI illness mediators at onset, at 6 weeks (on completion of the medication regimen) and 4 months after baseline; using 20 GWI patients. The response during and after an exercise challenge will be assessed followed by map the homeostatic networks in play over the 24 hours post-exercise in subjects before treatment, after completing the second treatment (week 6) and 4 months after initiating treatment (week 16).

ELIGIBILITY:
Inclusion Criteria:

* Male Veterans who were deployed in 1990 -1991 Gulf War.
* Veterans who currently meet the Kansas Gulf War Study Case Definition for Gulf War Illness.
* Veterans who were in good health based on medical history prior to 1990.
* Veterans who are between 40 to 70 years old
* Veterans who currently do not have exclusionary diagnoses that could reasonably explain the symptoms of their fatiguing illness and their severity.

Exclusion Criteria:

* Major depression with psychotic or melancholic features
* Schizophrenia
* Bipolar disorder
* Delusional disorders
* Dementias of any type
* History or current alcohol abuse
* History or current drug abuse
* Organ failure
* Transplant
* Defined rheumatologic
* Inflammatory disorders
* HIV
* Hepatitis B and C
* Primary sleep disorders
* Steroids
* Immunosuppressives
* Medications that impact immune function such as Enbrel or Methotrexate
* Tuberculosis or past history of tuberculosis exposure, as documented by PPD positivity

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker response to therapy using Cytokine panel | Change from Baseline at 6 weeks and 16 weeks
  Goal is decreased inflammation

SECONDARY OUTCOMES:
Biomarker response too therapy using VO2 exercise test | Change from Baseline at 6 weeks and 16 weeks]
  Goal is that both will prove safe for use in GWI patients

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Klimas, MD, Principal Investigator — South Florida Veterans Affairs Foundation for Research and Education
Locations (1):
- Miami VA Healthcare System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided